CLINICAL TRIAL: NCT03919487
Title: Correlation Between Surrogate Quality Indicators for Adenoma Detection Rate (ADR) and Adenoma Miss Rate (AMR) in Qualified Colonoscopy: CORE Study
Brief Title: Surrogate Quality Indicators for Adenoma Detection Rate (ADR)
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Gun, Kim. M.D., Ph.D., Professor, Soonchunhyang University Hospital
Other Study IDs: CORE study
Record Dates: First submitted 2019-03-07; First posted 2019-04-18 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Colon Adenoma
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Back-to-back colonoscopy group: As I described the study method in the protocol, the experimental group will be a screening colonoscopy cohort with back to back method. In fact, this study is to evaluate the correlation between quality indicators of colonoscopy and adenoma miss rate (AMR), and intervention is a single arm for back-to-back colonoscopy.
  Interventions: Procedure: Back to back colonoscopy

INTERVENTIONS:
Procedure: Back to back colonoscopy — After first colonoscopy performing with polypectomy, the 2nd colonoscopy will be performed right after the 1st colonoscopy, and if the missed lesion during the 1st colonoscopy will be found, it should be removed.
  Other Names: colonoscopy

SUMMARY:
This study is to evaluate the correlation of adenoma missing rate and quality indicators of colonoscopy including adenoma detection ratee (ADR), polyp detection rate (PDR), adenoma per colonoscopy rate (APC), adenoma per positive participant (APP), ADR-Plus, and to find out the surrogate indicators of ADR. This study is a prospective observational multi-center study. Correlation between AMR and quality indicators of colonoscopy based on the previous studies, 8 endoscopists participated in this study and will enroll 50 screening colonoscopies respectively.

Recruit research participants who want to participate in research in outpatient clinics. Perform colonoscopy in the morning after colon cleansing with split method. Colonoscopy is performed by back-to-back two consecutive colonoscopies. When the first colonoscopy is performed, the colonoscope is retracted after inserting the cecum, and all colon polyps are removed. After retracting to the anus of the first colonoscopy, the second colonoscopy is performed immediately. In case of newly detected colon polyps except for the small polyps and S-colon and rectal polyps which were left as photographs during the first colonoscopy with the second colonoscopy, we regard them as an overlooked lesion during the first colonoscopy. After the procedure, the histologic examination is confirmed and classified as benign lesions (all adenomas, advanced adenomas, dysplasia, and colorectal cancer) and non-lesion lesions.

Using the back-to-back colonoscopy results of the participants during the study period, calculate the quality indicators including ADR, PDR, APC, ADR-plus, APP and AMR for each endoscopist. And then, evaluate the correlation between AMR and other quality indicators.

DETAILED DESCRIPTION:
Background Colonoscopy reduces the risk of colorectal cancer by 77% and reduces mortality from colorectal cancer by more than 30%. However, in spite of the advantages of colonoscopy, the meta-analysis reported an incidence of intermediate cancer of 3.7%. In the case of proximal colon, the incidence of intermediate cancer was 2.4 times higher than that of the distal colon.

There are several possible causes of intermediate cancers, such as missed lesion during the previous colonoscopy, early-growth tumors before the follow-up period, and incomplete resection of the lesions. About 70-80% intermediate cancers are known to be originated from an missed lesion on endoscopy, and 10 ~ 27% is known to be caused by incomplete resection of the lesion on the previous colonoscopy.

The quality of colonoscopy for the prevention of intermediate cancer was first reported by the American Society of Gastrointestinal Endoscopy (ASGE) / American College of Gastroenterology (ACG) Task Force on Quality in Endoscopy in 2006 and the recently revised Quality indicators for colonoscopy (Quality index of colonoscopy) '.

The most popular and practically being used quality indicator of colonoscopy is an adenoma detection rate (ADR).

ADR is calculated as the number of colonoscopy with ≥1 adenoma detected during the colonoscopy divided by the total number of colonoscopies. ACGTF recommended the criteria of the quality index of the colonoscopy prior to the revision ADR was defined as 25% or more for men and 15% or more for women.

However, a Polish study reported a 10-fold higher risk of intermediate cancer when ADR was below 20%, and a recent large study by Corley showed that the incidence of colorectal cancer could be reduced by 3% and the mortality rate of colorectal cancer by 5% or more, especially when the ADR is increased by 1%.

Based on the evidence that the higher the ADR and the lower the risk of colorectal cancer, the quality index of colonoscopy was revised in 2015. Currently, the recommended ADR is 30% for men and 20% for women.

Although ADR appears to be a perfect quality marker, it requires a diagnosis of adenoma of the pathologic outcome in order to obtain ADR.

In particular, the calculation of ADR is based on the assumption that more than one adenoma is diagnosed during colonoscopy. However, even if the number of adenomas diagnosed during colonoscopy is different for each endoscopist, the concept of ADR does not distinguish this difference.

In fact, many recent studies have reported that endoscopist with an ADR more than 40% showed more than 20% adenoma missing rate.

The recent proposed measures to replace ADR include polyp detection rate (PDR) and adenoma per colonoscopy rate (APC). As with ADR, PDR is a measure of the rate at which more than one colorectal polyps are found in a colonoscopy practitioner aged 50 years or older. Unlike ADR, PDR does not need pathologic result. Recently, several studies have been reported that PDR can replace ADR and can be correlated with colorectal cancer prevention. The APC is different from that of ADR, and it is considered to be one of the alternative indicators that can compensate the shortcomings of "one and done" concept of ADR, because it can reflect the number of all adenomas found in the entire colon. According to a single-institution study using more than 20,000 colonoscopy analyzes that the recommended values for ADR 20% for men and women with ADR 15% for men over 50 years of age were APC 0.3.

In addition to APC, Adenoma per positive participants (APP), the total number of adenomas of participants divided by the number of examinees of adenomas detected (positive APPs), and the number of ADR-plus (ADR-plus) in the average number of additional found adenomas per test case divided by total colonoscopy were also introduced as quality indicators to predict the overlook of the lesion substitute for ADR.

In this regard, various substitute factors such as PDR, APC, and recently reported APP and ADR-plus have been introduced as an index parameter that can be used as a quality index to reflect the neglect of adenomas during colonoscopy. However, there is a very limited study of the direct comparison of correlation between each quality indicators and adenoma miss rate (AMR), and also the investigators have very limited knowledge which quaility incidator can well reflect the AMR.

The aim of this study was to investigate the efficacy of quality indicators which could best reflect the AMR and to find surrogate markers of ADR.

The primary endpoint of this study is to evaluate the relationship between known quality markers such as ADR, PDR, APC, APP, ADR-Plus, and AMR is examined.

This study will be performed as a cross-sectional study with prospective design.

Total of eight expert colonoscopists will participate in this study, and collecting the 50 colonoscopy data in each endoscopist. All enrolled cases will be subject for screening colonoscopy aged 50-75 years old.

This study excluded the colonoscopy cases with inappropriate bowel preparation, inflammatory bowel disease patients, and high-risk patients with family history of hereditary colorectal cancer.

Colon cleansing will be performed by the split method. Colonoscopy is performed by back-to-back two colonoscopies. When the first colonoscopy is performed, the colonoscope is retracted after inserting the cecum, and all colon polyps are removed. Only small polyps less than 5 mm located in the S-colon and rectum are left after photographing.

After performing the first colonoscopy, the second colonoscopy is performed immediately. A newly founded polyp (except polypoid and S-colon and rectal polyp which was left as a photograph at the time of 1st colonoscopy when performing a second colonoscopy) will be considered as a missed lesion and will be removed. After the procedure, confirm the presence of adenomatous polyps by pathologic results and record them on the case record. Using the back-to-back colonoscopy results of the participants during the study period, calculate the quality indicators including ADR, PDR, APC, ADR-plus, APP, and AMR. The correlations between ADR, PDR, APC, ADR-plus, APP, and AMR are compared using Pearson correlation constants.

ELIGIBILITY:
Inclusion Criteria:

* A 50-to 75-year-old colon cancer screening colonoscopist who has had previous colonoscopy experience or has had a colonoscopy within the last 5 years

Exclusion Criteria:

1. Total bowel preparation deficient (total bowel preparation by Boston bowel preparation scale <6 or any region score <2)
2. Inflammatory bowel disease patients
3. Family history of hereditary colorectal cancer (family history of two or more colorectal cancer or family history of at least one cancer diagnosed before age 60)
4. History of colorectal cancer or colon surgery
5. If the insertion of the appendix fails
6. A patient who does not agree with sleep induction calming

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community based, screening colonoscopy subjects
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Correlation between adenoma missing rate during the colonoscopy and other colonoscopy quality indicators in each endoscopist. | Within 1 year
  colonoscopy quality indicators including adenoma detection rate, polyp detection rate, adenoma per colonoscopy, adenoma detection rate-plus, adenoma per positive participant

SECONDARY OUTCOMES:
Evaluation of surrogate indicators of ADR | Within 1 year
  Correlation between ADR and other substitute indicators including PDR, APC, ADR-P

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Gun Kim, Professor, Study Director — Soonchunhyang University College of Medicine
Locations (1):
- Soonchunhyang univerisity hospital, Seoul, South Korea